CLINICAL TRIAL: NCT02941107
Title: The ORVAC Trial: A Phase IV, Double-blind, Randomised, Placebo-controlled Clinical Trial of a Third Scheduled Dose of RV1 Rotavirus Vaccine in Australian Indigenous Infants to Improve Protection Against Gastroenteritis
Brief Title: Optimising Rotavirus Vaccine in Aboriginal Children
Acronym: ORVAC
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Telethon Kids Institute (Other)
Collaborators: Menzies School of Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVID/2015-03
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Viral Gastroenteritis Due to Rotavirus
Keywords: Aboriginal; Rotavirus; Vaccine; Diarrhoea
MeSH Terms: conditions — Diarrhea | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotarix (Experimental): Rotarix (RV1) vaccine, 1mL liquid suspension administered orally.
  Interventions: Drug: Rotarix (RV1)
- Placebo (Placebo Comparator): Placebo liquid suspension manufactured to mimic Rotarix (RV1) vaccine, 1ml administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotarix (RV1) — ROTARIX™ (RV1) is a live-attenuated human monovalent oral vaccine containing attenuated G1P[8] human rotavirus strain sponsored and distributed in Australia by GlaxoSmithKline Biologicals where it is licensed for the prevention of rotavirus gastroenteritis.
  Other Names: ROTARIX™
  Arms: Rotarix
Drug: Placebo — The placebo for this trial will be Viscosweet, a clear and flavoured solution used as a pharmaceutical excipient repackaged into a labelled syringe identical to the active and firmly sealed with an end cap.
  Other Names: Viscosweet
  Arms: Placebo

SUMMARY:
Australian Indigenous children, particularly those living in remote communities, suffer a disproportionately high burden of rotavirus gastroenteritis disease. Despite the introduction of rotavirus vaccine into the Northern Territory (NT) Immunisation Schedule in 2006, the rate of hospitalization for rotavirus in NT Aboriginal children < 5 years continues to be high, and the rate ratio of rotavirus hospitalisations for Indigenous versus non-Indigenous children has actually increased. The reasons for sub-optimal vaccine response are not completely understood, but both reduced vaccine immune responses and low vaccine coverage are likely to be important factors.

The purpose of this study is to determine if Aboriginal children who receive an additional dose of RV1 between the ages of 6 and 12 months, will have an increase anti-rotavirus serum IgA seroconversion and decreased medical presentations with gastroenteritis in the first three years of life, compared to those who receive placebo.

DETAILED DESCRIPTION:
Australian Indigenous children, particularly those living in remote communities, suffer a disproportionately high burden of rotavirus gastroenteritis disease. Despite the introduction of rotavirus vaccine into the Northern Territory (NT) Immunisation Schedule in 2006, the rate of hospitalization for rotavirus in NT Aboriginal children < 5 years continues to be high, and the rate ratio of rotavirus hospitalisations for Indigenous versus non-Indigenous children has actually increased. The reasons for sub-optimal vaccine response are not completely understood, but both reduced vaccine immune responses and low vaccine coverage are likely to be important factors.

This study will enrol Aboriginal infants aged 6 months to < 12 months old who have received one or two prior doses of RV1. The coprimary aim is to determine whether an oral dose of RV1 vaccine at age 6 months to less than 12 months, compared to placebo, results in an increase in the average time to medical attendance for gastroenteritis before age 36 months (co-primary endpoint 1), and/ or superior immune protection against rotavirus gastroenteritis assessed approximately 1 to 2 months after vaccination (co-primary endpoint 2), in Australian Indigenous children.

This is a phase IV, randomised, placebo-controlled Bayesian trial with two strata representing residency based on a standard geographical classification of remoteness. It has the following key features:

1. Double-blind, randomised, placebo-controlled trial;
2. The procedures for enrolment, intervention, end-point and analysis are based on the principles of pragmatic trial design;
3. Non-fixed sample size up to 1,000 participants based on Bayesian stopping rules;
4. Fixed 1:1 enrolment into the active and control arm throughout the trial;
5. Frequent interim analyses can result in the trial stopping early for futility or expected success.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 6 months and < 12 months
* Identified as Aboriginal and/or Torres Strait Islander and/or South Sea Islander per attending legally responsible care-giver/parent.
* Have received either one or two prior doses of RV1 vaccination as confirmed by checking the immunisation register.
* Legally responsible care-giver/parent is willing for their infant to participate in the study and is aware of the requirements of the protocol.
* Legally responsible care-giver/parent is willing to allow other parties involved in the treatment of their child (including general practitioner, medical centre staff and any other medical professionals the child may be a patient of for the duration of the trial) to be notified of their participation in the trial and for participation in the trial to be recorded within the Northern Territory Immunisation Register.
* The legally responsible care-giver/parent is willing to allow the study team to obtain a vaccination history from Northern Territory Immunisation Register and/or the Australian Childhood Immunisation Register (ACIR) and/or local provider.
* The legally responsible care-giver/parent is willing to allow the study team to obtain a medical history from hospitalisation and laboratory databases, the disease notification register, the participant's electronic medical records and/or from the participant's primary care provider for the period from enrolment to age 36 months
* Informed consent for the infant's/child's participation in the study has been given by the legally responsible care-giver/parent

Exclusion Criteria:

Has any contraindication for RV1 vaccination including:

* Severe combined immunodeficiency, any history of intussusception, any history of hypersensitivity to any vaccine component, or an uncorrected gastrointestinal tract malformation, receipt of more than two weeks of immunosuppressant or immune modifying drugs, (e.g. prednisolone > 0.5mg/kg/day) within 28 days of enrolment, confirmed or suspected severe immunosuppressive or immunodeficient conditions, including human immunodeficiency virus (HIV) infection
* Receipt of any rotavirus vaccination other than RV1
* Receipt in the previous 3 months of any blood products including immunoglobulin
* Has received no prior doses or > two prior doses of RV1 vaccination
* Medical condition or treatment with medication which in the opinion of the clinic staff would make the child unsuitable for the trial
* Previously enrolled in the trial

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time from randomisation to medical attendance for acute gastroenteritis or acute diarrhoea illness | Randomisation to 36 months
  Time from randomisation to medical attendance (hospitalisation, emergency department presentation, medical clinic presentation) for which the primary reason for presentation is presumed or confirmed acute gastroenteritis or acute diarrhoea illness between randomisation and age 36 months.
Occurrence of anti-rotavirus IgA seroconversion | 28-55 Days post RV1/placebo administration
  Anti-rotavirus IgA seroconversion, defined as serum anti-rotavirus IgA > 20U/ ml 28 to 55 days post RV1/placebo among infants with anti-rotavirus serum IgA < 20U/ ml before RV1/placebo, to be summarised as the proportion of all children per group.

SECONDARY OUTCOMES:
Time from randomisation to hospitalisation for acute gastroenteritis or acute diarrhoea illness | Randomisation to 36 months
  Time from randomisation to hospitalisation for which the primary coded reason for admission is presumed or confirmed acute gastroenteritis or acute diarrhoea illness between randomisation and age 36 months.
Time from randomisation to hospitalisation for rotavirus confirmed diarrhoea illness | Randomisation to 36 months
  Time from randomisation to hospitalisation for which rotavirus confirmed diarrhoea illness occurs between randomisation and age 36 months.
Time from randomisation to Rotavirus infection | Randomisation to 36 months
  Time from randomisation to rotavirus infection meeting the jurisdictional case definition between randomisation and age 36 months.
Change in anti-rotavirus IgA log titre between administration of intervention (RV1/placebo) and 28 to 55 days post dose | Randomisation and 28-55 days post RV1/placebo administration
  Change in anti-rotavirus IgA log titre between administration of intervention (RV1/placebo) and 28 to 55 days post dose, to be summarised as the proportion of all children per group.
Occurrence of intussusception fulfilling Brighton criteria (see Appendix A) | Within the first 28 days of RV1/placebo administration
  The occurrence of intussusception fulfilling Brighton criteria (see Appendix A) within the first 28 days after RV1/placebo administration, to be summarised as the proportion of all children per group.
Occurrence of a serious adverse event | Randomisation to 36 months
  Serious adverse events between randomisation and age 36 months, to be summarised as the proportion of all children per group.
Medical attendance for confirmed acute gastroenteritis or acute diarrhoea illness between randomisation and 36 months gastroenteritis or acute diarrhoea illness. | Randomisation to 36 months
  Medical attendance (hospitalisation, emergency department presentations, medical clinic presentations) from the time of randomisation to age 36 months, for which the primary reason for presentation is presumed or confirmed acute gastroenteritis or acute diarrhoea illness, to be summarised as the proportion of all children per group.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Snelling, Principal Investigator — Telethon Kids Institute
Locations (1):
- Menzies School of Health Research, Darwin, Northern Territory, Australia

IPD SHARING:
Plan to Share IPD: Yes
IPD (de-identified) may be shared with other research teams subject to approval of the statistical analysis plan, data transfer agreement and appropriate ethics. However, prior approvals may be required from lead ethics
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: post publication of study results
Access Criteria: Researchers need to supply a statistical analysis plan and appropriate Ethics approvals

REFERENCES:
- [Derived] Middleton BF, Danchin M, Jones MA, Leach AJ, Cunliffe N, Kirkwood CD, Carapetis J, Gallagher S, Kirkham LA, Granland C, McNeal M, Marsh JA, Waddington CS, Snelling TL. Immunogenicity of a Third Scheduled Dose of Rotarix in Australian Indigenous Infants: A Phase IV, Double-blind, Randomized, Placebo-Controlled Clinical Trial. J Infect Dis. 2022 Nov 1;226(9):1537-1544. doi: 10.1093/infdis/jiac038. PMID 35134951
- [Derived] Jones MA, Graves T, Middleton B, Totterdell J, Snelling TL, Marsh JA. The ORVAC trial: a phase IV, double-blind, randomised, placebo-controlled clinical trial of a third scheduled dose of Rotarix rotavirus vaccine in Australian Indigenous infants to improve protection against gastroenteritis: a statistical analysis plan. Trials. 2020 Aug 26;21(1):741. doi: 10.1186/s13063-020-04602-w. PMID 32843086
- [Derived] Middleton BF, Jones MA, Waddington CS, Danchin M, McCallum C, Gallagher S, Leach AJ, Andrews R, Kirkwood C, Cunliffe N, Carapetis J, Marsh JA, Snelling T. The ORVAC trial protocol: a phase IV, double-blind, randomised, placebo-controlled clinical trial of a third scheduled dose of Rotarix rotavirus vaccine in Australian Indigenous infants to improve protection against gastroenteritis. BMJ Open. 2019 Nov 14;9(11):e032549. doi: 10.1136/bmjopen-2019-032549. PMID 31727664